CLINICAL TRIAL: NCT01488929
Title: A Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Study to Assess Efficacy, Safety, and Tolerability of TC-5619 as Augmentation Therapy to Improve Negative Symptoms and Cognition in Outpatients With Schizophrenia
Brief Title: Efficacy, Safety, and Tolerability of TC-5619 as Augmentation Therapy to Improve Negative Symptoms and Cognition in Outpatients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-5619-23-CRD-003
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia; Negative Symptoms; Cognitive Dysfunction
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — N-(2-(pyridin-3-ylmethyl)-1-azabicyclo(2.2.2)oct-3-yl)-1-benzofuran-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg TC-5619 (Experimental): One tablet of 5 mg TC-5619 will be administered orally once a day.
  Interventions: Drug: TC-5619
- 50 mg TC-5619 (Experimental): One tablet of 50 mg TC-5619 will be administered orally once a day.
  Interventions: Drug: TC-5619
- Placebo (Placebo Comparator): One tablet of placebo will be administered orally once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5619
  Arms: 5 mg TC-5619; 50 mg TC-5619
Drug: Placebo
  Arms: Placebo

SUMMARY:
Negative symptoms and cognitive dysfunction in schizophrenia (CDS) are core features of schizophrenia. These negative symptoms and cognitive deficits have a devastating impact on the function, employment, and social interactions of patients with schizophrenia. Medications used to treat schizophrenia (e.g. atypical antipsychotics) do not improve negative symptoms or CDS. TC-5619 is being developed for use as an add-on therapy in combination with atypical antipsychotics to treat patients with negative symptoms and CDS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia, per DSM-IV-TR criteria, as aided by the MINI International Neuropsychiatric Interview
2. Controlled schizophrenia, on stable dose of an approved atypical antipsychotic for at least 2 months prior to screening. Approved refers to regulatory approval in the country of use.
3. Stable schizophrenia as documented by lack of psychiatric hospitalization for 2 months prior to Screening (social admissions for the convenience of the subject allowed)
4. Clinical history of stable psychotic symptoms for 1 month prior to Screening.
5. Stable positive symptoms of schizophrenia for 4 weeks prior to Day 1, as shown by score ≤ 4 on PANSS for items related to delusion, hallucination, conceptual disorganization, and unusual thought content, at Screening and at Day 1.
6. Sum > 20 for the 7 items in the Negative Symptoms subscale of the PANSS.
7. Calgary Depression Schizophrenia Scale (CDSS) score < 6.
8. Simpson Angus Scale score < 12.
9. Outpatient with stable housing, and significant presence of an informant who is not a group home resident.

Exclusion Criteria:

1. Diagnosis of schizoaffective or schizophreniform disorders within 1 year prior to Screening.
2. Significant risk of suicide or attempted suicide in the 12 months before screening, or of danger to themselves or others.
3. Change in dosing of atypical antipsychotic within 2 months of Screening.
4. Treatment with electroconvulsive therapy (ECT) within 12 months of Screening.
5. Treatment with mood stabilizers, antidepressants, anxiolytics (short-acting hypnotics permitted), anticholinergics, or more than 1 antipsychotic within 1 month prior to Screening.
6. Treatment within 1 month prior to Screening with cognition-affecting agents other than the above (e.g. CNS stimulants).
7. History within past 6 months of screening of alcohol or illicit drug abuse.
8. Use of smoking cessation therapy within 1 month prior to Screening.
9. Positive urine drug screen except when related to prescribed short-acting benzodiazepines and opiates recently prescribed for an episode of acute pain (e.g., dental extraction).
10. History of significant other major or unstable neurological, neurosurgical (e.g. head trauma), metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disorder.
11. History of myocardial infarction based on medical history or electrocardiogram (ECG) findings at screening.
12. History of seizure disorder.
13. Type 1 diabetes mellitus.
14. Type 2 diabetes mellitus that requires medication (diet-controlled allowed, with HbA1C < 7.3).
15. Body Mass Index (BMI) > 35.
16. Uncontrolled hypothyroidism, vitamin B12 or folic acid deficiency.
17. Current TB or known systemic infection (e.g., HBV, HCV, HIV).
18. Clinically significant lab or ECG abnormality that could be a safety issue in the study, including QTcF > 450 for males and >470 for females.
19. Men, or women of child-bearing potential, who are unwilling or unable to use accepted methods of birth control as specified in Section 4.4.4
20. Women with a positive pregnancy test, or who are lactating.
21. Participated in another clinical trial within 3 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Scale for Assessment of Negative Symptoms (SANS) | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in the Cogstate Schizophrenia Battery (CSB) | 24 weeks
Change from baseline in UCSD Performance Based Skills Assessment, brief version (UPSA-Brief) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David P Walling, PhD, Principal Investigator — Collaborative Neuroscience Network, Inc
Locations (64):
- United States (22):
  - Collaborative Neuroscience Network, Inc, Garden Grove, California
  - Behavorial Research Specialists, Glendale, California
  - Apostle Clinical Trials, Inc, Long Beach, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Inc., Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - CNRI, San Diego, California
  - Segal Institute for Clinical Research, Lauderhill, Florida
  - Compass Research, LLC, Leesburg, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Precise Research Group, Flowood, Mississippi
  - St. Charles Psychiatric Associates - Midwest Reserch Group, Saint Charles, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - CRI Worldwide, LLC, Marlton, New Jersey
  - Behavioral Medical Research, Brooklyn, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Neuro-Behavorial Clinic Research, Inc., Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
- Hungary (5):
  - Semmelweis University, Department of Psychiatry, Budapest
  - University of Debrecen, Medical and Health Science Centre, Department of Psychiatry, Debrecen
  - Pharma4Trial Kft., Gyöngyös
  - University of Pecs, Department of Psychiatry, Pécs
  - St. George Hospital, Department of Psychiatry, Székesfehérvár
- Romania (5):
  - County Emergency Clinical Hospital of Arad, Arad, Arad
  - CMDTA Neomed, Brasov, Brașov County
  - Neuropsychiatry Clinical Hospital Craiova, Psychiatry Department, Craiova, Dolj
  - SC Lorentina 2102 SRL, Târgovişte, Dâmbovița County
  - University Emergency Central Military Hospital, Dept. of Psychiatry, Bucharest
- Russia (14):
  - Kemerovo Regional Clinical Psychiatric Hospital, Kemerovo
  - Moscow Research Institute of Psychiatry, Moscow
  - Menthal Health Research Center of the RAMS, Moscow
  - Nizhniy Novgorod Regional Psychoneurological Hospital # 1, Nizhny Novgorod
  - Saint-Petersburg State Public Healthcare Institution (City Psychiatric Hospital #7), Saint Petersburg
  - Saint-Petersburg State Public Healthcare Institution (Saint Nicholas Psychiatric Hospital), Saint Petersburg
  - Saint-Petersburg State Public Healthcare Institution (City Psychiatric Hospital #4), Saint Petersburg
  - Saint-Petersburg Research Psychoneurogical Institute, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution (City Psychiatric Hospital #6), Saint Petersburg
  - Municiple Healthcare Institution (City Clinical Hospital #2), Saratov
  - Institution of Russian Academy of Medical Sciences, Tomsk
  - Nizhny Novgorod Region State Budgetary Institution of Healthcare "Clinical Psychiatric Hospital #1 of Nizhny Novgorod", Veliky Novgorod
  - Yaroslavl State Medical Academy, Department of Psychiatry, Yaroslavl
  - Regional State Healthcare Institution (Sverdlovsk Regional Clinical Psychiatric Hospital), Yekaterinburg
- Serbia (6):
  - Clinical Centre "Dr Dragisa Misovic", Clinic of Psychiatry, Belgrade
  - Clinical Centre of Serbia, Clinic of Psychiatry, Belgrade
  - Institute of Mental Health, Belgrade
  - Clinical Centre Nis, Psychiatric Clinic, Gornja Toponica
  - Clinical Centre Kragujevac, Psychiatric Clinic, Kragujevac
  - Special Hospital for Psychiatric Diseases "Sveti Vracevi", Vojvodina
- Ukraine (12):
  - Crimean State Medical University (Dept. of Psychiatry), Simferopol, Autonomous Republic of Crimea
  - Odesa Regional Psychiatric Hospital #2, Odesa, Kominternivskyy District
  - Dnipropetrovsk Regional Clinical Hospital, Dnipropetrovsk
  - Dnipropetrovsk State Medical Academy, Dept. of Psychiatry, Dnipropetrovsk
  - Donetsk National Medical University (Regional Clinical Psychiatric Hospital), Donetsk
  - Institute of Neurology, Psychiatry and Narcology AMS of Ukraine, Kharkiv
  - Kharkiv Regional Clinical Psychiatric Hospital N 3, Kharkiv
  - Kyiv Station Railway Clinical Hospital # 1 of the STBA "South-Western Railway", Kyiv
  - Lugansk State Medical University, Luhansk
  - Odesa Regional Psychoneurological Dispensary, Odesa
  - Ukrainian Medical Stomatological Academy, Dept. of Psychiatry, Poltava
  - Vinnytsya National Medical University, Dept. of Psychiatry & Narcology, Vinnytsia